CLINICAL TRIAL: NCT00118326
Title: Feasibility of Granulocyte-Colony Stimulating Factor (G-CSF) Stimulated Bone Marrow From Pediatric Donors as a Stem Cell Source for Allogeneic Bone Marrow Transplant
Brief Title: Donor Bone Marrow Transplant in Treating Young Patients With Cancer or a Non-Cancerous Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Purpose: Treatment
Other Study IDs: 1802.00; FHCRC-1802.00; PBMTC-STC0233; CDR0000430709 (Registry Identifier: PDQ)
Record Dates: First submitted 2005-07-08; First posted 2005-07-11 (Estimated); Last update posted 2010-05-14 (Estimated); Status verified 2010-05

CONDITIONS: Kidney Cancer; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neuroblastoma; Sarcoma
Keywords: de novo myelodysplastic syndromes; disseminated neuroblastoma; previously treated myelodysplastic syndromes; recurrent neuroblastoma; secondary myelodysplastic syndromes; childhood acute myeloid leukemia in remission; childhood acute lymphoblastic leukemia in remission; childhood chronic myelogenous leukemia; juvenile myelomonocytic leukemia; previously treated childhood rhabdomyosarcoma; recurrent Wilms tumor and other childhood kidney tumors; recurrent/refractory childhood Hodgkin lymphoma; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood rhabdomyosarcoma; recurrent childhood small noncleaved cell lymphoma; untreated childhood acute lymphoblastic leukemia; untreated childhood acute myeloid leukemia and other myeloid malignancies
MeSH Terms: conditions — Kidney Neoplasms; Leukemia; Lymphoma; Myelodysplastic Syndromes; Neuroblastoma; Sarcoma; Leukemia, Myelomonocytic, Juvenile; Wilms Tumor; Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma | interventions — Filgrastim

INTERVENTIONS:
Biological: filgrastim
Procedure: allogeneic bone marrow transplantation

SUMMARY:
RATIONALE: A bone marrow transplant from a brother or sister may be able to replace blood-forming cells that were destroyed by chemotherapy or radiation therapy. Colony-stimulating factors, such as G-CSF, cause the body to make blood cells. Giving G-CSF to the donor may help the body make more stem cells that can be collected for bone marrow transplant and may cause fewer side effects in the patient after the transplant.

PURPOSE: This phase I/II trial is studying the side effects of donor bone marrow transplant and to see how well it works in treating young patients with cancer or a non-cancerous disease.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and feasibility of filgrastim (G-CSF)-mobilized bone marrow from an HLA-identical pediatric sibling donor as a stem cell source for pediatric patients undergoing allogeneic bone marrow transplantation for malignant or non-malignant disease.

Secondary

* Determine the time to neutrophil and platelet engraftment, number of red blood cell and platelet transfusions, number of febrile days, and number of hospitalization days in patients treated with this regimen.
* Determine the number of nucleated cells and CD34-positive cells, absolute lymphocyte count, and lymphocyte subsets (CD3/CD4/CD8) in G-CSF-mobilized bone marrow from these donors.

OUTLINE: This is a multicenter, pilot study.

Donors receive filgrastim (G-CSF) subcutaneously once daily on days -4 to 0. Donors then undergo standard bone marrow harvest on day 0.

Patients receive pre-transplantation conditioning and graft-versus-host disease prophylaxis according to the disease for which the patient is being treated and the treatment plan or clinical trial for which the patient is enrolled on. Patients undergo allogeneic bone marrow transplantation on day 0.

After completion of bone marrow harvest, donors are followed at 7 and 30 days. After completion of study treatment, patients are followed for 100 days post-transplantation and then periodically thereafter.

PROJECTED ACCRUAL: A total of 80 participants (40 donors and 40 patients) will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Patients (recipients):

  * Undergoing a myeloablative or nonmyeloablative allogeneic bone marrow transplantation for 1 of the following diseases:

    * Hematologic malignancy
    * Non-hematologic malignancy
    * Non-malignant disease
  * Not undergoing T-cell depleted bone marrow transplantation
* Donors:

  * Healthy sibling of a patient meeting eligibility requirements for this protocol
  * HLA-identically matched with patient

PATIENT CHARACTERISTICS:

Age

* 18 and under (patient and donor)

Performance status

* Karnofsky 90-100% (donor) OR
* Lansky 90-100% (donor)

Life expectancy

* Not specified

Hematopoietic

* No sickle cell anemia (donor)

Hepatic

* Not specified

Renal

* Not specified

Immunologic

* HIV negative (patient and donor)
* No uncontrolled bacterial, viral, fungal, or parasitic infection (donor)
* No potentially life threatening autoimmune disease (donor)

Other

* Not pregnant or nursing (patient and donor)
* Fertile patients must use effective contraception (patient)
* No other illness that would severely limit life expectancy (patient)
* No pre-existing medical condition that would confer a high risk for bone marrow donation (donor)
* No medical condition or psychiatric trait that would preclude G-CSF administration or bone marrow harvesting (donor)

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 years since prior allogeneic blood transfusion (donor)
* No concurrent growth factors post-transplantation (donor)

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* Concurrent participation in another treatment clinical trial allowed provided the use of filgrastim (G-CSF)-mobilized bone marrow is not excluded (patient)
* No other concurrent investigational agents (donor)

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2003-08; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety and feasibility

CONTACTS AND LOCATIONS:
Overall Officials: Ann E. Woolfrey, MD, Principal Investigator — Fred Hutchinson Cancer Center
Locations (2):
- United States (2):
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Fred Hutchinson Cancer Research Center, Seattle, Washington